CLINICAL TRIAL: NCT06965309
Title: Dose-escalation Study to Assess the Safety, Tolerability, and Preliminary Efficacy of HN2301 in Patients With Refractory Myasthenia Gravis (MG)
Brief Title: Efficacy and Safety of HN2301 in Refractory Myasthenia Gravis(MG)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Change of registrant
Sponsor: Shenzhen MagicRNA Biotechnology Co., Ltd (Industry)
Collaborators: Shanghai General Hospital (Songjiang Branch) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HN2301-002
Record Dates: First submitted 2025-04-29; First posted 2025-05-11 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Refractory Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HN2301 treatment group (Experimental): Specified dose level
  Interventions: Drug: HN2301 injection

INTERVENTIONS:
Drug: HN2301 injection — Description: Three dose groups were set up, starting from the low dose group and climbing to explore the safe and effective dose.
  Other Names: in vivo cart

SUMMARY:
This is an investigator-initiated trial designed to evaluate the safety, and efficacy of HN2301 in refractory myasthenia gravis

DETAILED DESCRIPTION:
This study is a prospective exploratory clinical trial in subjects with refractory myasthenia gravis. The objective is to evaluate the safety, initial efficacy of HN2301injection in refractory myasthenia gravis.

ELIGIBILITY:
Inclusion Criteria

* Age: 18-80 years, no gender restriction;
* Confirmed diagnosis of generalized myasthenia gravis (MG) with positive AchR or MuSK antibodies, meeting at least one of the following conditions:

  (1) Repetitive nerve stimulation suggesting neuromuscular transmission defect; (2) Positive response to neostigmine test; (3) Clinically judged improvement of --MG symptoms after oral cholinesterase inhibitor therapy;
* Clinical classification of MG according to MGFA types IIa-IVb (including IIa, IIb, IIIa, IIIb, IVa, IVb);
* Baseline MG-ADL (Myasthenia Gravis Activities of Daily Living) score ≥6, with ocular-related score <50%;
* Poor response and/or lack of effective treatment under standard therapies, defined as no improvement or worsening of symptoms despite stable treatment with corticosteroids, immunosuppressants (e.g., azathioprine, mycophenolate mofetil, tacrolimus, cyclosporin A, cyclophosphamide), or rituximab;
* Expected survival time greater than 12 weeks;
* Adequate bone marrow, coagulation, cardiopulmonary, liver, and renal function；Bone marrow function: ANC ≥1.5×10⁹/L, ALC ≥0.8×10⁹/L, Hb ≥80g/L; transfusions or growth factors must not be used within 7 days prior to screening to meet these criteria.Coagulation function: INR or APTT ≤1.5×ULN.
* Cardiac function: left ventricular ejection fraction (LVEF) ≥40% assessed by echocardiogram (ECHO).
* Pulmonary function: CTCAE grade ≤1 dyspnea and room air SpO₂ ≥92% (measured by pulse oximetry).
* Liver function: ALT and AST ≤2.5×ULN; total bilirubin <2.0 mg/dL (or <3.0 mg/dL for subjects with Gilbert's syndrome).
* Renal function: calculated creatinine clearance (Cockcroft-Gault) ≥50 mL/min without hydration assistance.

Exclusion Criteria

* Subjects positive for hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb) with detectable or quantifiable HBV DNA, positive for hepatitis C antibody (HCV Ab) with detectable or quantifiable HCV RNA, positive for HIV antibody, positive CMV DNA, or CMV DNA above the upper limit of detection; positive for syphilis antigen or antibody;
* Presence of other uncontrolled active infections;
* History of major organ transplantation (e.g., heart, lung, liver, kidney) or bone marrow/hematopoietic stem cell transplantation;
* Pregnant or breastfeeding women;
* Receipt of any mRNA-LNP products or other LNP-based drugs within the past two years;
* History of any of the following cardiovascular conditions within 6 months prior to screening: New York Heart Association (NYHA) Class III or IV heart failure, myocardial infarction, unstable angina, uncontrolled or symptomatic atrial arrhythmias, any ventricular arrhythmias, or other clinically significant cardiac disease;
* History of ≥Grade 2 bleeding events within 30 days prior to screening, or requiring long-term continuous anticoagulation therapy (e.g., warfarin, low molecular weight heparin, Xa factor inhibitors);
* History of live vaccination within 30 days prior to screening;
* Severe central nervous system diseases or pathological changes, including but not limited to: cerebrovascular accident, aneurysm, epilepsy, seizures/convulsions, aphasia, stroke, severe brain injury, dementia, Parkinson's disease, cerebellar disorders, organic brain syndromes, or psychosis;
* History of asthma or severe allergies;
* Any condition that, in the investigator's opinion, may increase the patient's risk or interfere with study assessments.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 9 (Actual)
Dates: Start 2026-01-19 (Actual); Primary Completion 2026-02-11 (Actual); Study Completion 2026-02-11 (Actual)

PRIMARY OUTCOMES:
Adverse events related to HN2301 | 3 months
  Incidence and severity of AEs associated with HN2301 as assessed by CTCAE v5.

SECONDARY OUTCOMES:
vivo CAR T cell production | Day-28 to14 days
  Assessment of CAR T production (CAR expression ratio in T cells) in the peripheral blood of MG patients by flow cytometry (FACS)
B cell ratio and counts in peripheral blood | Day-28 to12 months
  Assessment of B cell ratio and counts (B cell counts per μl peripheral blood) and B cell subsets(naive B cell, memory B cell) by flow cytometry (FACS) in peripheral blood
Change from baseline of MG-ADL score after HN2301 administration. | Day-28 to12 months
  1. Assessment of MG-ADL score from baseline administration at various timepoints up to month 12 follow-up visit. A total score can fall between 0 and 24 with a higher score representing a more significant degree of disease activity.
  2. Proportion of patients achieving a ≥2-point reduction in MG-ADL score following HN2301 administration.
Change from baseline of MGC score after HN2301 administration. | Day-28 to12 months
  1. Assessment of MGC score from baseline administration at various timepoints up to month 12 follow-up visit. A total score can fall between 0 and 50 with a higher score representing a more significant degree of disease activity.
  2. Proportion of patients achieving a ≥3-point reduction in MGC score following HN2301 administration.
Change from baseline of QMG score after HN2301 administration. | Day-28 to12 months
  1. Assessment of QMG from baseline administration at various timepoints up to month 12 follow-up visit. A total score can fall between 0 and 32, with a higher score representing a more significant degree of disease activity.
  2. Proportion of patients achieving a ≥3-point reduction in QMG score following HN2301 administration.
Change from baseline of MG-QOL15r score after HN2301 administration. | Day-28 to12 months
  Assessment of MG-QOL15r from baseline administration at various timepoints up to month 12 follow-up visit. A total score can fall between 0 and 100, with a lower score representing a more significant degree of disease activity.
Change of patients after HN2301 administration. | Day-28 to12 months
  1. Proportion of patients without symptom worsening
  2. Proportion of patients without symptom relapse
  3. Proportion of patients achieving minimal clinical manifestations
  4. Proportion of patients undergoing corticosteroid dose reduction
Time to achieve a ≥2 point reduction in MG-ADL score following HN2301 administration. | 14 days-12 months
  The time (months) to achieve a ≥2 point reduction in MG-ADL score following HN2301 administration of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Ailian Du, Principal Investigator — Shanghai Songshan Hospital
Locations (1):
- Shanghai General Hospital (Songjiang Branch) of Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No